CLINICAL TRIAL: NCT07160517
Title: Effectiveness of an Artificial Intelligence-Enabled Electric Toothbrush and Visual Pedagogy Materials on Oral Hygiene of Children With Autism Spectrum Disorder
Brief Title: AI Toothbrush and Visual Pedagogy to Improve Oral Hygiene in Children With Autism Spectrum Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marília Goulardins, PhD Candidate in Pediatric Dentistry, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CAAE80167324500005419
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Child; Oral Health; Artificial Intelligence
Keywords: Autism Spectrum Disorder, Toothbrushing, Oral Hygiene, Artificial Intelligence.
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: participants are randomized into two parallel arms: manual toothbrushing with visual pedagogy vs. AI-enabled electric toothbrush.
Masking Description: No masking will be applied. Both participants and investigators will be aware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Toothbrushing + Visual Pedagogy (Active Comparator): Participants will use a manual toothbrush with caregiver support. Visual pedagogy materials will be provided, including printed picture exchange communication system (PECS) cards illustrating each step of toothbrushing and tactile sensory panels simulating toothbrush bristles, toothpaste texture, and dental floss. Caregivers will be instructed to use these materials daily to improve comprehension and adherence to toothbrushing routines.
  Interventions: Behavioral: Visual Pedagogy and Manual Toothbrushing
- AI-enabled Electric Toothbrush (Experimental): Participants will use an Oral-B Genius X electric toothbrush equipped with artificial intelligence and Bluetooth connectivity. The device monitors brushing time, sequence, and pressure, providing real-time feedback through a smartphone application. Caregivers will be trained to supervise and encourage daily use at home for 3 weeks. The intervention aims to improve plaque removal and promote autonomy and motivation during oral hygiene in children with ASD.
  Interventions: Behavioral: Visual Pedagogy and Manual Toothbrushing

INTERVENTIONS:
Behavioral: Visual Pedagogy and Manual Toothbrushing — Participants in this arm will use a manual toothbrush with caregiver support. Visual pedagogy resources will include printed PECS cards illustrating each step of toothbrushing and tactile sensory panels simulating toothbrush bristles, toothpaste texture, and dental floss. Caregivers will be instructed to use these materials daily at home for 3 weeks to improve comprehension, adherence, and cooperation in children with ASD.
  Other Names: Visual support materials, Picture Exchange Communication System (PECS), tactile sensory panels

SUMMARY:
This randomized clinical trial evaluates the effectiveness of an AI-enabled electric toothbrush and visual pedagogy materials in improving oral hygiene among children with autism spectrum disorder (ASD). The study compares plaque control, gingival health, and adherence between children using a manual toothbrush with visual pedagogy support and those using an AI-enabled electric toothbrush with app-based monitoring.

DETAILED DESCRIPTION:
: Children with autism spectrum disorder (ASD) often face behavioral, motor, and sensory challenges that compromise their ability to perform effective toothbrushing. Caregivers are typically responsible for daily oral hygiene, yet few accessible digital or AI-based tools exist to support this process.

This study addresses this gap by combining two innovative approaches: visual pedagogy resources (picture exchange communication cards and tactile sensory panels) and an AI-enabled electric toothbrush with app-based monitoring. A randomized, parallel clinical trial will be conducted at the School of Dentistry of Ribeirão Preto, University of São Paulo (FORP-USP), including 60 children aged 6-12 years with ASD. Participants will be randomized into two groups:

* Group 1: Manual toothbrushing with caregiver support and visual pedagogy materials.
* Group 2: AI-enabled electric toothbrush (Oral-B Genius X) with app-based feedback monitoring brushing time, pressure, and sequence.

ELIGIBILITY:
Inclusion Criteria:Children aged 5-13 years with a prior diagnosis of autism spectrum disorder (ASD) level 1 , 2 or 3 confirmed by a neuropediatrician.

Child must be accompanied by a primary caregiver (≥18 years old) responsible for daily oral hygiene.

Caregiver must have access to a smartphone or computer to interact with the digital platform.

Written informed consent (TCLE) from the caregiver and assent (TALE) from the child.

-

Exclusion Criteria:Severe systemic medical conditions that contraindicate participation in clinical oral evaluations.

Children with advanced periodontal disease or other oral conditions requiring urgent dental treatment.

Caregivers who are unable or unwilling to use basic digital platforms (smartphone, tablet, or computer).

Families who decline participation at any stage of the study.

-

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in Plaque Index (Simplified Oral Hygiene Index - Greene & Vermillion) | Baseline, Week 3, Week 6
  Difference in gingival health between baseline and follow-up, assessed using the Löe and Silness Gingival Index. Higher scores indicate worse gingival condition.

SECONDARY OUTCOMES:
Bleeding on Probing (Community Periodontal Index) | Baseline, Week 6
  Assessment of bleeding on probing at six index teeth sites, following WHO Community Periodontal Index criteria.

OTHER OUTCOMES:
Caregiver-Reported Adherence and Motivation | Baseline, Week 6
  Questionnaire responses evaluating caregiver perceptions of the child's motivation, autonomy, and adherence to oral hygiene routines.
Usability of Digital Platform (System Usability Scale - SUS) | After 3 weeks of use
  Usability and acceptability of the caregiver support digital platform, assessed by the 10-item System Usability Scale (SUS). Scores range from 0 to 100; scores above 68 indicate good usability.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Nelson Filho, DDS, PhD, Study Director — Full Professor, Department of Pediatric Dentistry, School of Dentistry of Ribeirão Preto - USP
Locations (1):
- School of Dentistry of Ribeirão Preto - University of São Paulo (FORP-USP), Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided